CLINICAL TRIAL: NCT03175081
Title: Intraperitoneal Local Anesthetic in Bariatric Surgery: A Double Blind-randomized Controlled Pilot Trial
Brief Title: Intraperitoneal Local Anesthetic in Bariatric Surgery Study (iLABS Study)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Tikfu Gee (Other)
Responsible Party: Sponsor-Investigator, Dr. Tikfu Gee, Senior lecturer/ consultant, Universiti Putra Malaysia
Organization: Universiti Putra Malaysia (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NMRR-17-284-33857
Record Dates: First submitted 2017-05-24; First posted 2017-06-05 (Actual); Last update posted 2021-01-25 (Actual); Status verified 2021-01

CONDITIONS: Overweight and Obesity; Bariatric Surgery Candidate
Keywords: Intraperitoneal local anesthetic; Ropivacaine; Postoperative pain; Bariatric surgery; Sleeve gastrectomy
MeSH Terms: conditions — Overweight; Obesity; Pain, Postoperative | interventions — Ropivacaine; Saline Solution; Control Groups

STUDY DESIGN:
Intervention Model Description: The study will involve two groups with equal allocation of patients in the test group (local anaesthesia) and control group (normal saline) by randomization. All patients who agree to participate in this study will be randomized into one of the study groups.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test group (Experimental): Patients will undergo elective laparoscopic sleeve gastrectomy with ropivacaine diluted in normal saline injected along the stomach region at the end of the surgical procedure.
  Interventions: Drug: Ropivacaine
- Control group (Experimental): Patients will undergo elective laparoscopic sleeve gastrectomy with only normal saline injected along the stomach region at the end of the surgical procedure.
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Ropivacaine — Patient undergo elective laparoscopic sleeve gastrectomy will receive 20mL of 150mg ropivacaine (0.75%) diluted in 180mL normal saline to be injected through a catheter along the greater curvature and left subdiaphragmatic region of the stomach at the end of the surgical procedure. After the surgery, the medical doctors or nurses in the ward that is not otherwise involved in this research will assess and record the pain score using visual analog scale (VAS) (0-10). The abdomen and shoulder tip pain intensity will be rated at two, four, six, eight, 24 and 48 hours postoperatively.
  Other Names: Test group
  Arms: Test group
Drug: Normal saline — Patient undergo elective laparoscopic sleeve gastrectomy will receive 200mL normal saline to be injected through a catheter along the greater curvature and left subdiaphragmatic region of the stomach at the end of the surgical procedure. After the surgery, the medical doctors or nurses in the ward that is not otherwise involved in this research will assess and record the pain score using visual analog scale (VAS) (0-10). The abdomen and shoulder tip pain intensity will be rated at two, four, six, eight, 24 and 48 hours postoperatively.
  Other Names: Control group
  Arms: Control group

SUMMARY:
Obesity is a metabolic disorder that has gradually become a prevalent public health problem and is becoming one of the leading causes of death and disability worldwide. The most efficacious therapy for morbid obesity today is bariatric surgery. Bariatric surgery increases life expectancy by correcting the comorbidities associated with obesity, improves the quality of life, and is associated with reduced morbidity and mortality. There is an increase application of laparoscopic procedures as it is considered to cause less pain than traditional open surgery, smaller incision, reduced blood loss and shorter postoperative stay, which cuts down on hospital cost. However, postoperative pain still exists causing unpleasant experience for the patient and at times causes a delayed discharge. Pain after bariatric surgery is a result of many mechanisms such as tissue injury, abdominal distention, local trauma of the stomach, chemical irritation of the peritoneum, and the pneumoperitoneum and this pain potentially can prolong hospital stay and lead to increased morbidity, and bariatric surgeons are striving to minimize the morbidity of current procedures to improve patient outcomes and this gave rise to the use of intraperitoneal local anesthetics (LA). It was found that the use of intraperitoneal LA in laparoscopic cholecystectomy is safe, and it results in a statistically significant reduction in early postoperative abdominal pain. Many studies were done to evaluate the efficacy of intraperitoneal LA in laparoscopic cholecystectomy, gynecologic procedures and appendectomy but to date there are limited studies done to evaluate the role of intraperitoneal LA in bariatric surgery. The aim of this study is to evaluate the effectiveness of intraperitoneal instillation of local ropivacaine on postoperative abdominal pain after laparoscopic sleeve gastrectomy (LSG). We hypothesized that the administration of intraperitoneal instillation of local ropivacaine would help reduce postoperative pain.

DETAILED DESCRIPTION:
Recruitment will be a double-blind, placebo-controlled randomized study in patients age 18 and above going for laparoscopic sleeve gastrectomy (LSG). The study will involve two groups with equal allocation of patients in the test group (local anaesthesia) and control group (normal saline) by randomization. All patient will need to be evaluated by our multidisciplinary team before randomization. Each patient going for an elective LSG will be informed regarding this research study, and the final decision will solely be made based on patients' willingness. All patients who agree to participate in this study will be randomized into one of the study groups. The patients will also be made aware that this is an experimental trial and both verbal and written informed consent will be taken before treatment. In addition, the patients will be informed regarding the use of the clinical and analytical data for publication purposes.

Patients will not be given access to the study data however they will be informed regarding their progress during every follow-up visit. All research data will be kept in our hard disk as well as our web-based storage (i-cloud and i-drive) for two years. Study data will be held even after the study period as there will still be a continuous follow-up with the patients for life. However, all patients' information obtained from this study will be kept and handled in a confidential manner, by applicable laws and regulations. When publishing or presenting the study results, the identity of patients will not be revealed without patient's expressed consent. Participants will also be covered under clinical trial insurance from the institution during the study period. In the case of emergency, all patients will be given the contact number of the investigator as the investigator are contactable throughout the day. This study will begin after receiving the approval of Medical Research & Ethics Committee, Ministry of Health Malaysia.

Computer generated randomization will be done using Interactive Web Response Technology. There will be equal chances for patients to be assigned to either one of the study groups. The result of the randomization will be kept in envelopes and viewed by the research assistant who did not otherwise participate in this study, were unknown to the investigators and the patients, and the answer will be contained in a set of sealed envelopes. After admitting the patient into the operating room and just before the surgery was done, the numbered envelope will be opened by the operating theater nurse and the card inside determined which group the patient would be placed. The operating theater nurse will then prepare either 20mL of 150mg ropivacaine in 180mL normal saline (for test group) or 200mL normal saline (for control group) using a standard syringe and the syringe will be given to the surgeon who then injects the solution through a catheter along the greater curvature and left subdiaphragmatic region of the stomach. The general anesthetic used for all patients will be a combination of 1gm IV Paracetamol, 40mg IV Parecoxib and IV Fentamyl prepared according to patient's adjusted body weight.

Patients will need to be admitted to the hospital one day before the scheduled surgery date. Participating patients that are allergic to local anesthetic ropivacaine will be excluded from this study. However, if patients have allergy due to the medication after surgery, anti-allergic medication will be administered to the patients upon investigation. After the surgery, the medical doctors or nurses in the ward that is not otherwise involved in this research will assess and record the pain score using visual analog scale (VAS) (0-10). A score of 0 means no pain, whereas a score of 10 equals the worst pain ever experienced. Post-operative pain will be rated on a VAS at rest and cough. The time of arrival in the postoperative recovery room will be defined as zero hours postoperatively. The patients will be asked about the location of pain, whether at the shoulder, incision sites, and/or inside the abdomen by the medical doctors or nurses. The abdomen and shoulder tip pain intensity will be rated at two, four, six, eight, 24 and 48 hours postoperatively. The analgesic requirement during the 48 hours after the surgery will also be noted by the medical doctor or nurses in the ward. The duration of patients' participation in the study will only be for two days postoperative. However, patients still need to come for follow-up after surgery. The standard follow-up includes a visit to the outpatient clinic at 1, 2, 3, 4 weeks after surgery, then 3, 6, 9, 12, 18, 24 months and after that, a life-long annual visit. Adverse events (eg. post-operative bleeding and stapler leak) will be monitored closely at 1, 2, 3, and 4 weeks after surgery. In any occurrence of an adverse event, it will be documented and reported within 14 days.

Sample Size Estimation The sample size was estimated with the help of PS software (power and sample size calculation software) 3.0.43 with a power of 80% and a significant level of 0.05. The estimation was based on Visual Analog Score (VAS) with assuming 50% of difference in mean postoperative pain score. The total estimated sample size is 22 patients in each arm for our study. However, with the inclusion of 20% drop out rate, the total number of patients needed for this study is 27 patients in each arm.

Data Analysis Statistical calculations will be performed using the standard statistical software package, IBM SPSS Statistics for Windows, Version 23.0. Armonk, NY: IBM Corp. All data will be expressed as mean values and standard deviation, with the exception of rescue analgesic treatment and the occurrence of shoulder tip pain that will be in percentages (%). Median and interquartile range (IQR) will be calculated for all not normally distributed continuous variables. Non-parametric tests such as Mann-Whitney U test and/orKruskall-Wallis test will be used for non-normal distribution of variables. Associations between qualitative variables will be determined by Chi-square test, Fisher's exact test and SAS Exact Contingency Table. In all statistical analyses, p-value of < 0.05 (95% confidence interval) was considered to be statistically significant.

Study Ethics Ethical clearance will be obtained from the Medical Research Ethic Committee of the Faculty of Medicine, Universiti Putra Malaysia and Kuala Lumpur General Hospital. This study will be submitted for National Medical Research Register (NMRR). Respondent consent will be obtained from each participant of study.

Conflict of Interest There is no conflict of interest among the investigators.

ELIGIBILITY:
Inclusion Criteria:

i. Patients age 18 years and above ii. Patients who can communicate in English or Malay iii. Patients undergoing elective laparoscopic sleeve gastrectomy iv. Able to give informed consent

Exclusion Criteria:

i. Patients age below 18 years ii. Patients are allergic to ropivacaine or local anaesthetic iii. Inability to informed consent iv. American Society of Anesthesiologists Classification > 3 v. Patients with chronic medical diseases (eg. Ischaemic heart disease, cardiac arrhythmias, cardiac failure) and chronic opioid treatment vi. Patients with previous foregut surgery including esophageal, gastric, liver, and pancreas resections

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2017-04-27 (Actual); Primary Completion 2018-02-27 (Actual); Study Completion 2018-04-27 (Actual)

PRIMARY OUTCOMES:
2 hours postoperative pain at rest | 2 hours after surgery
  Measured by visual analogue pain scale
4 hours postoperative pain at rest | 4 hours after surgery
  Measured by visual analogue pain scale
6 hours postoperative pain at rest | 6 hours after surgery
  Measured by visual analogue pain scale
8 hours postoperative pain at rest | 8 hours after surgery
  Measured by visual analogue pain scale
24 hours postoperative pain at rest | 24 hours after surgery
  Measured by visual analogue pain scale
48 hours postoperative pain at rest | 48 hours after surgery
  Measured by visual analogue pain scale

SECONDARY OUTCOMES:
2 hours postoperative pain at cough | 2 hours after surgery
  Measured by visual analogue pain scale
4 hours postoperative pain at cough | 4 hours after surgery
  Measured by visual analogue pain scale
6 hours postoperative pain at cough | 6 hours after surgery
  Measured by visual analogue pain scale
8 hours postoperative pain at cough | 8 hours after surgery
  Measured by visual analogue pain scale
24 hours postoperative pain at cough | 24 hours after surgery
  Measured by visual analogue pain scale
48 hours postoperative pain at cough | 48 hours after surgery
  Measured by visual analogue pain scale

CONTACTS AND LOCATIONS:
Overall Officials: Lim Shu Yu, MS, Principal Investigator — Universiti Putra Malaysia
Locations (2):
- Malaysia (2):
  - Hospital Kuala Lumpur, Kuala Lumpur, Kuala Lumpur
  - Hospital Serdang, Kajang, Selangor

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sjostrom L. Bariatric surgery and reduction in morbidity and mortality: experiences from the SOS study. Int J Obes (Lond). 2008 Dec;32 Suppl 7:S93-7. doi: 10.1038/ijo.2008.244. PMID 19136998
- [Background] Lee YC, Lee CK, Liew PL, Lin YC, Lee WJ. Evaluation of quality of life and impact of personality in Chinese obese patients following laparoscopic sleeve gastrectomy. Hepatogastroenterology. 2011 Jul-Aug;58(109):1248-51. doi: 10.5754/hge10619. PMID 21937388
- [Background] Rosenthal RJ; International Sleeve Gastrectomy Expert Panel; Diaz AA, Arvidsson D, Baker RS, Basso N, Bellanger D, Boza C, El Mourad H, France M, Gagner M, Galvao-Neto M, Higa KD, Himpens J, Hutchinson CM, Jacobs M, Jorgensen JO, Jossart G, Lakdawala M, Nguyen NT, Nocca D, Prager G, Pomp A, Ramos AC, Rosenthal RJ, Shah S, Vix M, Wittgrove A, Zundel N. International Sleeve Gastrectomy Expert Panel Consensus Statement: best practice guidelines based on experience of >12,000 cases. Surg Obes Relat Dis. 2012 Jan-Feb;8(1):8-19. doi: 10.1016/j.soard.2011.10.019. Epub 2011 Nov 10. PMID 22248433
- [Background] Dixon JB, le Roux CW, Rubino F, Zimmet P. Bariatric surgery for type 2 diabetes. Lancet. 2012 Jun 16;379(9833):2300-11. doi: 10.1016/S0140-6736(12)60401-2. Epub 2012 Jun 9. PMID 22683132
- [Background] Wills VL, Hunt DR. Pain after laparoscopic cholecystectomy. Br J Surg. 2000 Mar;87(3):273-84. doi: 10.1046/j.1365-2168.2000.01374.x. PMID 10718794
- [Background] Parikh M, Issa R, McCrillis A, Saunders JK, Ude-Welcome A, Gagner M. Surgical strategies that may decrease leak after laparoscopic sleeve gastrectomy: a systematic review and meta-analysis of 9991 cases. Ann Surg. 2013 Feb;257(2):231-7. doi: 10.1097/SLA.0b013e31826cc714. PMID 23023201
- [Background] Pequignot A, Fuks D, Verhaeghe P, Dhahri A, Brehant O, Bartoli E, Delcenserie R, Yzet T, Regimbeau JM. Is there a place for pigtail drains in the management of gastric leaks after laparoscopic sleeve gastrectomy? Obes Surg. 2012 May;22(5):712-20. doi: 10.1007/s11695-012-0597-0. PMID 22328096
- [Background] Kim TH, Kang H, Hong JH, Park JS, Baek CW, Kim JY, Jung YH, Kim HK. Intraperitoneal and intravenous lidocaine for effective pain relief after laparoscopic appendectomy: a prospective, randomized, double-blind, placebo-controlled study. Surg Endosc. 2011 Oct;25(10):3183-90. doi: 10.1007/s00464-011-1684-3. Epub 2011 Apr 13. PMID 21487863
- [Background] Chazelet C, Verhaeghe P, Perterli R, Fennich S, Houdart R, Topart R, Tussiot J, Skawinski P, Seraille G, Catheline JM, Merabet M, Dehaye B, Pautot V, Juglard G, Sala JJ. [Longitudinal sleeve gastrectomy as a stand-alone bariatric procedure: Results of a multicenter retrospective study]. J Chir (Paris). 2009 Aug;146(4):368-72. doi: 10.1016/j.jchir.2009.08.021. Epub 2009 Sep 16. French. PMID 19762021
- [Background] Louizos AA, Hadzilia SJ, Leandros E, Kouroukli IK, Georgiou LG, Bramis JP. Postoperative pain relief after laparoscopic cholecystectomy: a placebo-controlled double-blind randomized trial of preincisional infiltration and intraperitoneal instillation of levobupivacaine 0.25%. Surg Endosc. 2005 Nov;19(11):1503-6. doi: 10.1007/s00464-005-3002-4. Epub 2005 Oct 3. PMID 16328673
- [Background] Elhakim M, Elkott M, Ali NM, Tahoun HM. Intraperitoneal lidocaine for postoperative pain after laparoscopy. Acta Anaesthesiol Scand. 2000 Mar;44(3):280-4. doi: 10.1034/j.1399-6576.2000.440310.x. PMID 10714840
- [Result] Barczynski M, Konturek A, Herman RM. Superiority of preemptive analgesia with intraperitoneal instillation of bupivacaine before rather than after the creation of pneumoperitoneum for laparoscopic cholecystectomy: a randomized, double-blind, placebo-controlled study. Surg Endosc. 2006 Jul;20(7):1088-93. doi: 10.1007/s00464-005-0458-1. Epub 2006 May 13. PMID 16703434
- [Result] Lepner U, Goroshina J, Samarutel J. Postoperative pain relief after laparoscopic cholecystectomy: a randomised prospective double-blind clinical trial. Scand J Surg. 2003;92(2):121-4. PMID 12841551
- [Result] Khan MR, Raza R, Zafar SN, Shamim F, Raza SA, Pal KM, Zafar H, Alvi R, Chawla T, Azmi R. Intraperitoneal lignocaine (lidocaine) versus bupivacaine after laparoscopic cholecystectomy: results of a randomized controlled trial. J Surg Res. 2012 Dec;178(2):662-9. doi: 10.1016/j.jss.2012.06.005. Epub 2012 Jun 22. PMID 22763212
- [Result] Malhotra N, Chanana C, Roy KK, Kumar S, Rewari V, Sharma JB. To compare the efficacy of two doses of intraperitoneal bupivacaine for pain relief after operative laparoscopy in gynecology. Arch Gynecol Obstet. 2007 Oct;276(4):323-6. doi: 10.1007/s00404-007-0337-1. Epub 2007 Jul 25. PMID 17653742
- [Result] Ceyhan T, Teksoz E, Gungor S, Goktolga U, Pabuccu R. Effect of bupivacaine after operative laparoscopic gynecologic procedures. J Minim Invasive Gynecol. 2005 Jul-Aug;12(4):326-9. doi: 10.1016/j.jmig.2005.05.003. PMID 16036192
- [Result] Jiranantarat V, Rushatamukayanunt W, Lert-akyamanee N, Sirijearanai R, Piromrat I, Suwannanonda P, Muangkasem J. Analgesic effect of intraperitoneal instillation of bupivacaine for postoperative laparoscopic cholecystectomy. J Med Assoc Thai. 2002 Sep;85 Suppl 3:S897-903. PMID 12452227
- [Result] Park YH, Kang H, Woo YC, Park SG, Baek CW, Jung YH, Kim JY, Koo GH, Kim SD, Park JS. The effect of intraperitoneal ropivacaine on pain after laparoscopic colectomy: a prospective randomized controlled trial. J Surg Res. 2011 Nov;171(1):94-100. doi: 10.1016/j.jss.2010.03.024. Epub 2010 Apr 8. PMID 20605604
- [Result] Ruiz-Tovar J, Gonzalez J, Garcia A, Cruz C, Rivas S, Jimenez M, Ferrigni C, Duran M. Intraperitoneal Ropivacaine Irrigation in Patients Undergoing Bariatric Surgery: a Prospective Randomized Clinical Trial. Obes Surg. 2016 Nov;26(11):2616-2621. doi: 10.1007/s11695-016-2142-z. PMID 27007272
- [Result] Lee IO, Kim SH, Kong MH, Lee MK, Kim NS, Choi YS, Lim SH. Pain after laparoscopic cholecystectomy: the effect and timing of incisional and intraperitoneal bupivacaine. Can J Anaesth. 2001 Jun;48(6):545-50. doi: 10.1007/BF03016830. PMID 11444448
- [Result] Symons JL, Kemmeter PR, Davis AT, Foote JA, Baker RS, Bettendorf MJ, Paulson JE. A double-blinded, prospective randomized controlled trial of intraperitoneal bupivacaine in laparoscopic Roux-en-Y gastric bypass. J Am Coll Surg. 2007 Mar;204(3):392-8. doi: 10.1016/j.jamcollsurg.2006.12.013. PMID 17324772